CLINICAL TRIAL: NCT02210767
Title: Effects of Walnuts on Central Blood Pressure, Arterial Stiffness Indices, Lipoproteins, and Other CVD Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PKE ALA
Record Dates: First submitted 2014-07-17; First posted 2014-08-07 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Walnut Diet (Experimental): Provides ~2 oz. walnuts/day (2-3% of total calories from alpha-linolenic acid [ALA])
  Interventions: Other: Walnut Diet
- Walnut Control Diet (Active Comparator): Provides same fatty acid profile (<7% SFA, 9% MUFA, 14-15% PUFA, 2-3% ALA) as Walnut Diet, but is devoid of walnuts and their bioactives
  Interventions: Other: Walnut Control Diet
- Low ALA Diet (Placebo Comparator): Provides similar macronutrient and linoleic acid profile but replaces ALA with oleic acid (<7% SFA, 12% MUFA, 12% PUFA, 0.5% ALA)
  Interventions: Other: Low ALA Diet

INTERVENTIONS:
Other: Walnut Diet — 2 oz. walnuts/day (2-3% of total calories from ALA)
  Arms: Walnut Diet
Other: Walnut Control Diet — 2-3% ALA but no walnuts provided
  Arms: Walnut Control Diet
Other: Low ALA Diet — ALA replaced by oleic acid
  Arms: Low ALA Diet

SUMMARY:
This study will evaluate the effects of walnut-derived ALA and bioactives on multiple CVD risk factors, including central blood pressure, arterial stiffness indices, inflammatory markers, urinary isoprostanes, vascular adhesion markers, and changes in lipids and lipoproteins. Gut microbiome changes due to walnut consumption will also be assessed using the 16S rRNA gene.

DETAILED DESCRIPTION:
Diets containing nuts likely reduce cardiovascular disease (CVD) risk but the mechanisms remain poorly defined. Walnuts contain substantial amounts of polyunsaturated fatty acids (PUFAs), particularly alpha-linolenic acid (ALA), and are a rich source of bioactives. Many vegetable oils are high in PUFAs but most lack ALA and do not provide the same complement of bioactive compounds as walnuts. ALA is thought to improve cardiovascular health by modulating circulating lipid concentrations, altering membrane structure/function by enhancing the total ω-3 fatty acid content of cell membrane phospholipids, and reducing inflammatory reactions by inhibiting production of arachidonic acid-derived eicosanoids. Consumption of walnuts has consistently been shown to improve blood lipids/lipoproteins and vascular health. However, there remains much debate over what is the preferable replacement for saturated fat in the diet. Because of the ALA and bioactives that they provide, walnuts may confer specific CVD benefits. To study the effects of walnuts, in terms of both their ALA content and bioactive compounds, we will compare two test diets (one containing walnuts and one matched for PUFA and ALA content but devoid of walnuts and their bioactives) to a control diet matched for macronutrient and linoleic acid (LA) content but providing oleic acid in place of ALA. This diet design will provide information about how walnuts affect the selected endpoints of interest due to their bioactives as well as their ALA content, and whether walnut ALA is a superior substitute for dietary saturated fat compared to oleic acid.

Feeding protocol and study treatments:

This study is designed as a double-blind, 3-period, randomized, cross-over controlled feeding study. Prior to randomization, participants will complete a two week run-in on a standard Western diet. Each diet period treatment phase will be 6 weeks in duration, separated by 2-week washout periods. The three test diets are: 1) a walnut diet (WD; providing ~2.0 oz of walnuts per day); 2) a matched walnut control diet (WCD) that will provide the same fatty acid profile as the walnut diet, but will not contain walnuts (and their bioactives); and 3) a low ALA diet (LAD) with a similar macronutrient (and linoleic acid) composition as the WD and WCD, but using oleic acid to replace ALA. Study diets will be prepared in a metabolic kitchen, with three isocaloric meals and a snack provided each day, based on a 7-day rotating menu cycle. Participants will be instructed to consume only the prepared foods and limit their intake of alcohol to 2 drinks/week and caffeinated calorie-free beverages to 40 ounces (5 drinks) per day. Diets will be planned for every subject according to his/her energy requirements and will be nutritionally adequate. This diet design will permit the WD to be compared with the WCD and LAD and, thereby, allow us to ascertain the specific effects that walnuts and their bioactive components (including and beyond ALA) may have on CVD risk factors and artery health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-65 years
* BMI greater than 25 and less than or equal to 40 kg/m2
* Non-smokers
* TG < 350 mg/dL
* LDL-C between the 25-95th percentile from NHANES:
* Males: 105-194 mg/dL
* Females: 98-190 mg/dL
* Stage I hypertension:
* SBP > 120 mmHg and/or DBP > 80 mmHg
* SBP < 160 mmHg and DBP < 100 mmHg
* Free of established CVD, stroke, diabetes, liver, kidney or autoimmune disease.

Exclusion Criteria:

* Elevated BP (SBP ≥160 mmHg OR DBP ≥ 100 mmHg)
* A history of myocardial infarction, stroke, diabetes mellitus, liver disease, inflammatory disease, kidney disease, and/or thyroid disease (unless controlled on medication).
* Blood pressure or cholesterol-lowering medication use
* Refusal to discontinue intake of putative cholesterol-lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, and phytoestrogens).
* Vegetarianism or other dietary practices that are inconsistent with the test diets
* Nut allergies (Other food allergies will be reviewed on a case-by-case basis)
* Refusal to discontinue nutritional supplements, herbs, vitamins or NSAID's
* Latex allergy
* Pregnant or lactating females

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in central blood pressure at the end of diet period 1 (week 6), end of diet period 2 (week 14), and end of diet period 3 (week 22) | End of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)

SECONDARY OUTCOMES:
Change in 24-hour ambulatory blood pressure | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in indices of arterial stiffness (pulse wave velocity) | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in lipoprotein particle size | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
  The VAP© Test provides a direct measure of the following lipid and lipoprotein classes and subclasses: LDL, Lp(a), IDL, LDL1, LDL2, LDL3, LDL4, HDL, HDL2, HDL3, VLDL, VLDL1+2, VLDL3, TC, TG, Non-HDL, Remnant Lipoproteins, ApoB100, and ApoA1
Change in inflammatory cytokines (tumor necrosis factor-alpha and interleukin-6) | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in the composition of the gut microbiome | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
  This will be assessed via sequencing of microbial 16S rRNA from fecal samples.
Change in serum C-reactive protein | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in serum glucose | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in serum insulin | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in urinary F2α-isoprostanes | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in lipid/lipoprotein profile | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides
Change in heart rate variability | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)
Change in vascular adhesion markers (VCAM and ICAM) | Week 0, end of diet period 1 (week 6), end of diet period 2 (week 14), end of diet period 3 (week 22)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Sabate J, Fraser GE, Burke K, Knutsen SF, Bennett H, Lindsted KD. Effects of walnuts on serum lipid levels and blood pressure in normal men. N Engl J Med. 1993 Mar 4;328(9):603-7. doi: 10.1056/NEJM199303043280902. PMID 8357360
- [Background] Zhao G, Etherton TD, Martin KR, West SG, Gillies PJ, Kris-Etherton PM. Dietary alpha-linolenic acid reduces inflammatory and lipid cardiovascular risk factors in hypercholesterolemic men and women. J Nutr. 2004 Nov;134(11):2991-7. doi: 10.1093/jn/134.11.2991. PMID 15514264
- [Background] Banel DK, Hu FB. Effects of walnut consumption on blood lipids and other cardiovascular risk factors: a meta-analysis and systematic review. Am J Clin Nutr. 2009 Jul;90(1):56-63. doi: 10.3945/ajcn.2009.27457. Epub 2009 May 20. PMID 19458020
- [Background] West SG, Krick AL, Klein LC, Zhao G, Wojtowicz TF, McGuiness M, Bagshaw DM, Wagner P, Ceballos RM, Holub BJ, Kris-Etherton PM. Effects of diets high in walnuts and flax oil on hemodynamic responses to stress and vascular endothelial function. J Am Coll Nutr. 2010 Dec;29(6):595-603. doi: 10.1080/07315724.2010.10719898. PMID 21677123
- [Background] Estruch R, Ros E, Salas-Salvadó J, Covas MI, Corella D, Arós F, Gómez-Gracia E, Ruiz-Gutiérrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L,Pintó X, Basora J, Muñoz MA, Sorlí JV, Martínez JA, Martínez-González MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013;368:1279-1290.
- [Background] Zhang J, Grieger JA, Kris-Etherton PM, Thompson JT, Gillies PJ, Fleming JA, Vanden Heuvel JP. Walnut oil increases cholesterol efflux through inhibition of stearoyl CoA desaturase 1 in THP-1 macrophage-derived foam cells. Nutr Metab (Lond). 2011 Aug 26;8:61. doi: 10.1186/1743-7075-8-61. PMID 21871057
- [Derived] Petersen KS, Chandra M, Chen See JR, Leister J, Jafari F, Tindall A, Kris-Etherton PM, Lamendella R. Walnut consumption and gut microbial metabolism: Results of an exploratory analysis from a randomized, crossover, controlled-feeding study. Clin Nutr. 2023 Nov;42(11):2258-2269. doi: 10.1016/j.clnu.2023.09.023. Epub 2023 Sep 28. PMID 37826992
- [Derived] Tindall AM, McLimans CJ, Petersen KS, Kris-Etherton PM, Lamendella R. Walnuts and Vegetable Oils Containing Oleic Acid Differentially Affect the Gut Microbiota and Associations with Cardiovascular Risk Factors: Follow-up of a Randomized, Controlled, Feeding Trial in Adults at Risk for Cardiovascular Disease. J Nutr. 2020 Apr 1;150(4):806-817. doi: 10.1093/jn/nxz289. PMID 31848609
- [Derived] Tindall AM, Petersen KS, Skulas-Ray AC, Richter CK, Proctor DN, Kris-Etherton PM. Replacing Saturated Fat With Walnuts or Vegetable Oils Improves Central Blood Pressure and Serum Lipids in Adults at Risk for Cardiovascular Disease: A Randomized Controlled-Feeding Trial. J Am Heart Assoc. 2019 May 7;8(9):e011512. doi: 10.1161/JAHA.118.011512. PMID 31039663